CLINICAL TRIAL: NCT00812890
Title: Exploring Semi-Quantitative Pregnancy Tests and Their Impact on Reproductive Health Service Provision
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Gynuity Health Projects (Other)
Responsible Party: Dr Paul D Blumenthal, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-11042008-1333; 14922
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

INTERVENTIONS:
Device: semi-quantitative pregnancy test

SUMMARY:
This study will examine the feasibility, practicality, utility and usability of a semi-quantitative urine pregnancy test (dBest One Step hCG Panel Test Kit) recently approved by the food and drug administration (FDA) for both Professional (physician office) and over-the-counter (consumer) use. The study seeks to:

1. Assess the correlation of this pregnancy test results with serum values (as distinct from urine) hCG.
2. Assess whether or not time of day of urine collection has any impact on the outcome of the dBest test.
3. Assess user comprehension of the pregnancy test, especially assessment of the result.

DETAILED DESCRIPTION:
This study will examine the feasibility, practicality, utility and usability of a semi-quantitative urine pregnancy test (dBest One Step hCG Panel Test Kit) recently approved by the food and drug administration (FDA) for both Professional (physician office) and over-the-counter (consumer) use. The study seeks to:

1. Assess the correlation of this pregnancy test results with serum values (as distinct from urine) hCG.
2. Assess whether or not time of day of urine collection has any impact on the outcome of the dBest test.
3. Assess user comprehension of the pregnancy test, especially assessment of the result.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older, presenting for early abortion, pre-natal care, or fertility services.
* If pregnant, gestational age < 84 days by LMP, ultrasound or clinical assessment.
* Agrees to return for follow-up visit and willing to provide an address and/or telephone number for purposes of follow-up.
* Able to consent to study participation.

Exclusion Criteria:

* Women less than 18 years of age.
* Women who are not pregnant, except if presenting for IVF services.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess the correlation between this pregnancy test's results with serum values (as distinct from urine) hCG. 2. To assess whether or not urine concentration has any impact on the outcome | 15 minutes pregnancy test reading

SECONDARY OUTCOMES:
To assess user comprehension of the test. | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Dr Paul D Blumenthal, Principal Investigator — Stanford University; Richard Fischer, Sub-Investigator — Planned Parenthood Mar Monte; Steve Lichtenberg, Sub-Investigator — Family Planning Associates Medical
Locations (3):
- United States (3):
  - Planned Parenthood Mar Monte, Sacromento, California
  - Stanford University School of Medicine, Stanford, California
  - Family Planning Associates Medical, Chicago, Illinois